CLINICAL TRIAL: NCT03947671
Title: Active Temperature Management After Cardiac Surgery and Its Effect on Postoperative Cognitive Dysfunction
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Loss of funds
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Stryker Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM20015426
Record Dates: First submitted 2019-04-25; First posted 2019-05-13 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Cardiac Surgery; Post-operative Cognitive Dysfunction; Fever
Keywords: temperature regulation
MeSH Terms: conditions — Fever | interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Body wrap (Experimental): This group will receive the body wraps post surgery to maintain normothermia.
  Interventions: Device: Rapr Rounds Hyper/Hypothermia Wraps
- Tylenol (Active Comparator): This group will receive the standard of care of monitoring temperature and administering Tylenol if a fever develops.
  Interventions: Drug: Acetaminophen
- Tylenol with body wrap (Experimental): This group will receive the standard of care of monitoring temperature but will be administered Tylenol and body wraps if a fever develops.
  Interventions: Device: Rapr Rounds Hyper/Hypothermia Wraps; Drug: Acetaminophen

INTERVENTIONS:
Device: Rapr Rounds Hyper/Hypothermia Wraps — Rapr Round® vest and leg wraps will placed around the torso and legs of the participant and will be adjusted to maintain normal body temperature
  Arms: Body wrap; Tylenol with body wrap
Drug: Acetaminophen — Acetaminophen will be administered as it would be per standard of care
  Other Names: Tylenol
  Arms: Tylenol; Tylenol with body wrap

SUMMARY:
This study will assess the effect of active postoperative temperature management and its effect on the cognitive function in patients following coronary artery bypass graft (CABG) surgery to determine if active postoperative temperature management to maintain normothermia reduces postoperative cognitive dysfunction (POCD) in this population. Additionally, the investigators will explore differences in temperature control variability by using temperature management wraps combined with acetaminophen vs. acetaminophen alone in a pilot arm.

DETAILED DESCRIPTION:
As one of the more common hospital-based major interventional procedures, 180,476 CABG surgeries were performed in the United States in 2016, according to the Society of Thoracic Surgeons Adult Cardiac Surgery Database (STS ACSD). Of these, 23,545 operations also involved aortic or mitral valve repair or replacement. The demographic characteristics of patients undergoing cardiac surgery have changed over time, with a higher proportion of elderly patients undergoing increasingly complex procedures. The number of patients with neurological disease prior to surgery has nearly doubled from 1.4% in 2001 to nearly 2.8% as of 2010, and is rising as surgical care improves and includes more such patients .

The recognition of neurological complications associated with cardiac surgery has been report-ed widely, and neurological dysfunction can be categorized as type 1 (brain death, non-fatal stroke, and new transient ischemic attack) or type 2 (delirium and postoperative cognitive dys-function) . The incidence postoperative neurological complications, defined as "permanent stroke" by the STS ACSD, was noted in 2016 to be 1.3% following isolated CABG operations, but was noted to be higher, between 2-3% in CABG patients also receiving aortic or mitral valve surgery as part of their operation. Notably, this statistic does not capture POCD, although steps are being taken to better capture this, perhaps as a patient-reported outcome (PRO) in the future.

As early as 1955, POCD was described by Bedford in the Lancet under the designation "adverse cerebral effects of anesthesia on old people" . It can affect any age group, but does seem to dis-proportionately affect patients age 60 or older, causing difficulty in daily life and their ability to return to work . Short-term POCD, up to 6 weeks postoperatively, occurs in 20-50% of patients undergoing cardiac surgery. Longer-term POCD, defined as a subtle deterioration in cognitive function 6 months following surgery, occurs in 10-30% of cardiac surgery patients . In a longitudinal study with 8.5 years of follow-up, Steinmetz et al. found POCD to be associated with higher mortality (Cox proportional hazard ratio 1.63, 95% confidence interval 1.11-2.38; p = 0.01), earlier retirement, and greater utilization of social financial assistance . Monk et al. found that the risk of death within one year was greater among patients who had POCD when they were discharged from the hospital .

CABG and valve surgery most commonly use the extracorporeal cardiopulmonary bypass machine to perfuse the body during cardiac surgery. The aorta is cross-clamped to allow work and suturing in a near bloodless field. The major blood branches to the brain come off the aorta. When the aorta is cross-clamped, the brain undergoes a period of ischemia. While the patient is on bypass, the body and brain are kept at low temperatures to quell the effects of ischemia. Temperature elevation has been proposed to have an all-or-none response with a defined threshold beyond which the increased temperature aggravates ischemic injury. Hyperthermia leads to physiological and structural changes in the brain which include alterations of enzyme activity and damage to cytoskeletal proteins found in the brain. In addition, hyperthermia causes a release of excitatory neurotransmitters, the production of free radicals, an increase in blood-brain barrier permeability, and increase in intracellular acidosis after ischemic reperfusion all of which have all been proposed as mechanisms through which hyperthermia leads to brain tissue injury and can exacerbate ischemic brain injury .

Intraoperative temperature during cardiac surgery has long been thought to have an association with postoperative neurological outcomes, and has been well studied. In mitigating neuroinflammation and subsequent brain injury, intraoperative hypothermia as compared with normothermia has been the subject of much debate, and outcomes have varied considerably in various studies. The process of rewarming patients as they gradually disengage from cardiopulmonary bypass has been noted as another important process in modulating neuroprotection, and has al-so been studied extensively. Nearly all studies have associated a slower rate of intraoperative rewarming with a decreased incidence of POCD.

Postoperative hyperthermia is a much less well-studied phenomenon. It occurs in approximately 30% of all CABG patients , and one study has associated it with POCD, noting that patients with supra-normal temperatures in the first 24-hour postoperative period following CABG have poorer cognitive outcomes when compared to those with normal temperatures in this setting .

At our institution and many others, the current standard of care pertaining to postoperative hyperthermia management in cardiac surgery patients involves treatment with acetaminophen and room temperature if it rises to greater than or equal to 38.3 degrees.

The Altrix Precision Temperature Management System, and specifically the Rapr Round® product, offers a means by which medical staff may be able to control temperature in cardiac surgery patients postoperatively, while preventing fever from occurring and in per our hypothesis, may be able to decrease short term POCD and its associated sequelae in this patient population. This temperature management system is intended for circulating temperature controlled warm or cold water via patient contact thermal transfer devices for the application of regulating human body temperature in situations where a physician or clinician with prescription privileges determines that temperature therapy is necessary or desirable.

For this study, the Rapr Round® vest and leg wraps are placed around the torso and legs of the patient and adjust body temperature by circulating water through channels in the wrap. In this case the wraps will be used to maintain patient temperature in the intervention group at 36.5 +/- 0.2 degrees Celsius, or normothermia.

ELIGIBILITY:
Inclusion Criteria:

1. scheduled coronary artery bypass graft surgery patients, with or without valve surgery
2. patients able to give informed consent

Exclusion Criteria:

1. age < 20 years or > 89 years
2. patients with unscheduled CABG +/- valve surgery (i.e. emergency surgery)
3. deformity or skin condition of chest or thighs that would interfere with the successful placement of Rapr Round® vest and leg wraps
4. patients presenting to the ICU postoperatively with a fever ≥ 38.3
5. patients with planned intraoperative circulatory arrest
6. prisoners
7. pregnant patients
8. patients with symptomatic cerebrovascular disease, specifically residual motor deficits, expressive or receptive aphasia from prior stroke or cerebrovascular accident

Ages: 20 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive Function post CABG | From pre surgery and 6 weeks post surgery
  Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) administered by a clinical psychologist or re-searcher specifically trained by the clinical psychologist. The RBANS is a screening tool that has been standardized to measure the neu-ropsychological status of adult patient between the ages of 20 and 89. It is composed of 12 sub-tests and takes approximately 30 minutes to administer. It is scored using a scaled index score from 40 to 160 with the following score ranges:
  130 and above: very superior 120-129: superior 110-119: high average 90-109: average 80-89: low average 70-79: borderline 69 and below: extremely low

SECONDARY OUTCOMES:
Variability in Temperature | Up to 24 hours post surgery
  Pattern of body temperature during post-op period measured using electronic thermometers

CONTACTS AND LOCATIONS:
Overall Officials: Vishal Yajnik, MD, MS, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No